CLINICAL TRIAL: NCT06875817
Title: Effects of Feldenkrais Exercises on Pain, Range of Motion, and Disability in Patients With Knee Osteoarthritis
Brief Title: Effects of Feldenkrais Exercises in Knee Osteoarthritis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0150
Record Dates: First submitted 2025-03-10; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis (Knee OA)
Keywords: Disability; Feldenkrais Method; Goniometry; Knee Osteoarthritis; Numeric Pain Rating Scale; Range of Motion
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-A (Feldenkrais exercises) (Experimental): This group of participants will engage in Feldenkrais exercises focused on pain, improved mobility, and disability. Each session will last 30 minutes, conducted twice a week for 4 weeks. The exercises include Pelvic Clock Exercise, Knee Rolling, Ankle Circles, Knee Flexion and Extension and Leg Slides.
  Interventions: Other: Feldenkrais exercises
- Group-B (Standard Physicaltherapy interventions) (Active Comparator): Participants will receive standard physical therapy interventions for knee osteoarthritis.
  Protocol:
  * Knee Isometrics: Isometric exercises targeting the quadriceps and hamstrings, performed for 10 minutes, twice a week.
  * Knee Mobilization
  * Transcutaneous Electric Nerve Stimulation (TENS).
  * Heating Pad Duration: 30-minute sessions, conducted twice a week for 4 weeks.
  Interventions: Other: Standard physical therapy interventions

INTERVENTIONS:
Other: Feldenkrais exercises — Feldenkrais exercises focused on pain, improving mobility, and disability.
  Arms: Group-A (Feldenkrais exercises)
Other: Standard physical therapy interventions — * Knee Isometrics: Isometric exercises targeting the quadriceps and hamstrings, performed for 10 minutes, twice a week.
  * Knee Mobilization
  * Transcutaneous Electric Nerve Stimulation (TENS).
  * Heating Pad Duration: 30-minute sessions, conducted twice a week for 4 weeks.
  Arms: Group-B (Standard Physicaltherapy interventions)

SUMMARY:
The primary objective of the study is to determine the effects of Feldenkrais Exercises on Pain, Range of Motion, and Disability in Patients with Knee osteoarthritis. Knee osteoarthritis poses significant challenges in pain management, mobility improvement, and disability reduction among middle-aged to older adults. Feldenkrais Method offers benefits comparable to back school lessons or core stability exercises. This study, conducted as a Randomized Controlled Trial at RIPHAH Rehabilitation Clinic, aims to assess the efficacy of Feldenkrais exercises compared to conventional physical therapy in addressing pain, range of motion, and disability in knee osteoarthritis patients aged 40-60 years. A non-probability convenience sampling method will recruit 32 participants meeting specific criteria for osteoarthritis severity and functional ability. Participants will be randomly assigned to Group A (Feldenkrais exercises) or Group B (conventional therapy), with interventions delivered over four weeks. Group A will engage in Feldenkrais exercises targeting pelvic and lower limb mobility, while Group B will receive standard treatments including knee isometrics, mobilization, transcutaneous electric nerve stimulation, and heating pad applications. Pain severity will be measured using the Numeric Pain Rating Scale, Range of Motion assessed via goniometry, and disability evaluated using the Western Ontario McMaster Universities Osteoarthritis Index. Statistical analysis using SPSS will compare outcomes between groups at baseline, post-treatment, and follow-up assessments.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is one of the most prevalent rheumatic diseases in the elderly, being a frequent cause of incapacity among this population. It is more common in the knee and is characterized by pain, stiffness, and function loss. OA is a major public health problem. The prevalence of knee OA is 34-45% in the Indian population with clinical symptoms of pain, reduced muscle strength, and knee function. That is the most common form of degenerative joint disease affecting 15 to 40% of people aged 40 and above. One hundred fifty-one million people worldwide experienced OA, and it was ranked sixth as a leading cause of moderate and severe disability. The knee is the joint most frequently affected by osteoarthritis. The Feldenkrais Method has the potential to help older people with OA. Developed by Dr. Moshe Feldenkrais, the method is a gentle form of exercise which has been shown to be acceptable for older people who have limited movement. The Feldenkrais Method is taught in two parallel forms, Awareness Through Movement (conducted as a group exercise) and Functional Integration (one-on one approach). This study explores the effectiveness of Awareness Through Movement lessons in helping older people with OA. The method aims for improved functioning, where the entire body cooperates efficiently with minimal effort. This study aims to explore the potential benefits of Feldenkrais exercises as an alternative, non-invasive treatment for knee osteoarthritis. Medical conventional treatments for knee OA, such as pharmacotherapy and surgical interventions, often come with limitations including potential side effects, high costs, and sometimes limited long-term effectiveness. These constraints necessitate the exploration of alternative, non-invasive treatment options that can be both effective and accessible. Feldenkrais exercises focus on improving movement patterns and body awareness, which may help reduce pain, enhance range of motion, and decrease disability.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 to 60 years of patients.
* Both female and male
* Able to walk for 6 minutes (Timed up-and-go test)
* Able to rise from floor
* Grade 2 and 3 of osteoarthritis diagnosed with radiograph (Kellgren and Lawrence classification system)
* Pain reported on VAS score ˃6/10 in knee region for more than 3 months

Exclusion Criteria:

* • Tuberculosis, carcinoma, heart disease, and osteoporosis

  * Any trauma or localized infection in the knee joint
  * Hyper flexibility
  * Open sores
  * Ongoing radiotherapy, chemotherapy, steroid therapy, or anticoagulants
  * Psychiatric diseases such as phobia/obsession and depression
  * Allergy to hot pack
  * Patients with a history of surgery in the knee region within a year.
  * Severe cognitive impairments
  * Contraindications to physical activity
  * Concurrent participation in other physical therapy programs

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-09-02 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | upto 4 weeks
  The NPRS is a segmented numeric scale in which the respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The common format is a horizontal bar or line. NPRS is anchored by terms describing pain severity extremes.
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | upto 4 weeks
  WOMAC is a disease-specific measure of health status (pain, stiffness, and function) in OA sufferers. It is widely used for evaluating hip and knee osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales
Universal Goniometer (UG) | upto 4 weeks
  A universal goniometer is a crucial tool in orthopedics used to precisely measure joint angles. It exists in two primary forms: the short-arm version is ideal for smaller joints such as the wrist, elbow, or ankle, while the long-arm version is more accurate for joints with longer levers like the knee and hip. It highlighting its role in quantifying joint mobility and aiding in treatment planning and assessment in medical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam Fatima, PhD*, Principal Investigator — Riphah International University
Locations (1):
- RIPHAH Rehabilitation Clinic, Punjab, Pakistan, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brooks PM. The burden of musculoskeletal disease--a global perspective. Clin Rheumatol. 2006 Nov;25(6):778-81. doi: 10.1007/s10067-006-0240-3. Epub 2006 Apr 12. PMID 16609823
- [Background] Zhang Y, Jordan JM. Epidemiology of osteoarthritis. Clin Geriatr Med. 2010 Aug;26(3):355-69. doi: 10.1016/j.cger.2010.03.001. PMID 20699159
- [Background] Vincent KR, Vincent HK. Resistance exercise for knee osteoarthritis. PM R. 2012 May;4(5 Suppl):S45-52. doi: 10.1016/j.pmrj.2012.01.019. PMID 22632702
- [Background] Salaffi F, Carotti M, Stancati A, Grassi W. Health-related quality of life in older adults with symptomatic hip and knee osteoarthritis: a comparison with matched healthy controls. Aging Clin Exp Res. 2005 Aug;17(4):255-63. doi: 10.1007/BF03324607. PMID 16285189
- [Background] Webb R, Cofre Lizama LE, Galea MP. Moving with ease: feldenkrais method classes for people with osteoarthritis. Evid Based Complement Alternat Med. 2013;2013:479142. doi: 10.1155/2013/479142. Epub 2013 Sep 3. PMID 24078825
- [Background] Lespasio MJ, Piuzzi NS, Husni ME, Muschler GF, Guarino A, Mont MA. Knee Osteoarthritis: A Primer. Perm J. 2017;21:16-183. doi: 10.7812/TPP/16-183. PMID 29035179